CLINICAL TRIAL: NCT03164811
Title: Goal Directed Fluid Therapy Based on Pulse Pressure Variation Compared With Standard Fluid Therapy in Patients Undergoing Complex Spine Surgery: a Randomized Controlled Trial
Brief Title: GDFT Based on PPV Compared With Standard Fluid Therapy in Patients Undergoing Complex Spine Surgery: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si826/2016
Record Dates: First submitted 2017-04-24; First posted 2017-05-24 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Spine Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDFT group (Experimental): The GDFT group will receive 400 ml of 12.5% carbohydrate drink after 6 pm until the bed time in the day before surgery and 200 ml in the morning of the surgery day. Acetate ringer solution will be start at 7:00. After induction PPV will be measure and fluid bolus 200 ml in 10 minutes will be given if PPV >13 before prone position. During the operation, the patient in GDFT group will receipt fluid therapy according to acceptable PPV
  Interventions: Procedure: goal directed fluid therapy
- controlled group (Other): The carbohydrate drink will not be given. Fluid, blood and blood product administration will be under attending anesthesiologist order.
  Interventions: Other: Controlled

INTERVENTIONS:
Procedure: goal directed fluid therapy — pulse pressure variation will be used to as a goal to guide fluid administration in this group
  Arms: GDFT group
Other: Controlled — standard fluid treatment by an anesthesiologist
  Arms: controlled group

SUMMARY:
The investigators will do the Goal directed fluid therapy by protocolized fluid management in the experimental group, using PPV to guide the fluid administration, compare with standard fluid management in patients undergoing complex spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* elective surgery
* thoracic/lumbar spine surgery >= 3 levels and duration >= 3 hours

Exclusion Criteria:

* Cr >2 mg/dl or eGFR < 60 ml/min
* coronary artery disease, congestive heart failure or cardiac arrhythmia
* BMI >30 kg/m2
* hemodynamic unstable, preoperatively
* uncontrolled hypertension
* respiratory system compliance < 30 ml/cmH2O

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
episode of intraoperative hypotension | intraoperative
  Blood pressure will be record continuously using arterial catheter in both group. Number of participants and episode of hypotension (defined as SBP < 90 mmHg or MAP < 60 mmHg or decrease of SPB >= 25% from baseline for 5 minutes or need vasopressor) therapy

SECONDARY OUTCOMES:
unit of blood transfusion | intraoperative and up to 24 hours postoperatively
  all unit of blood transfusion will be record intraoperative and postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No